CLINICAL TRIAL: NCT04289246
Title: Supporting the Medication Adherence of Older Mexican Adults Through External Cues Provided With Ambient Displays: Protocol of a Feasibility Randomized Controlled Trial
Brief Title: Supporting the Medication Adherence of Older Mexican Adults Through External Cues Provided With Ambient Displays
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autonoma de Baja California (Other)
Responsible Party: Principal Investigator, Marcela D. Rodriguez, Full Time Professor, Universidad Autonoma de Baja California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 105/6/C/103/18
Record Dates: First submitted 2020-02-11; First posted 2020-02-28 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Medication Adherence; Medication Compliance
Keywords: older adult; frail elderly; mobile health
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Intervention Model Description: The study included baseline, intervention, and postintervention phases. Half of the participants were randomly allocated to the treatment group (n=8), and the other half was assigned to the control group (n=8). During the study phases, research assistants measured medication adherence weekly through the pill counting technique.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (TG) (Experimental): On the first day of the intervention phase, research assistants visited TG's participants to introduce the MAD in the presence of caregivers. After the training session, which lasted 40 min approximately, the MAD was personalized according to the participant's prescriptions and through discussions with them on an appropriate schedule for presenting the reminders. Research assistants used the MAD administrator sub-system to enter the medication names, health problems to address, timetables, and the frequency at which medications should be taken. Then, they attached and configured NFC tags to each of the pill containers, which included selecting the images that best represented the pills and their containers to be used to form the visual reminders. Afterward, the MAD was placed in the homes' area where participants reported taking medications. MAD was used for 5 weeks during which data on medication adherence and system adoption was collected from the TG.
  Interventions: Device: Medication Ambient Display (MAD)
- Control Group (CG) (No Intervention): Participants in the CG followed their medication routine as usual. During 5 weeks data on medication adherence was collected.

INTERVENTIONS:
Device: Medication Ambient Display (MAD) — MAD was implemented for Android tablets to provide the following external cues:
  * Abstract and stylized representations of medication adherence. The MAD shows a virtual birdcage, which has the aim of raising elders' consciousness about how they have to take responsibility for caring for their health, in a way similar to willingly caring for a pet. Each day, a newborn pet grows to represent medication compliance. By touching any point on the parakeet's virtual cage, the MAD presents information on the participants' daily medication compliance.
  * Auditory and visual reminders. The parakeet provides auditory reminders (a parakeet whistle) and pictograms to inform the medication to take.
  After participants take their medication, they move the MAD closer to the pill container to indicate that the medication was taken. This functionality was implemented through Near Field Communication (NFC) technology. Afterward, the parakeet acknowledges that the medication was registered as taken.
  Arms: Treatment Group (TG)

SUMMARY:
Background: Problems with prospective memory, which refer to the ability to remember future intentions, cause deficits in basic and instrumental activities of daily living, such as taking medications. Older adults show minimal deficits when they rely on mostly preserved and relatively automatic associative retrieval processes. On the basis of this, the investigators of this study propose to provide external cues to support the automatic retrieval of an intended action, that is, to take medicines. To reach this end, the Medication Ambient Display (MAD) was developed. It is a system that unobtrusively presents relevant information unless it requires the users' attention, It uses different abstract modalities to provide external cues that enable older adults to easily take their medications on time and be aware of their medication adherence.

Objective: This study aimed to assess the adoption and effect of external cues provided through MAD on medication adherence in older adults. The study aimed to address the following research questions:

1. What is the effect of the external cues provided by the MAD on older adults' medication adherence?
2. How do the MAD design features promote its adoption?

Methods: A total of 16 older adults, who took at least three medications and had mild cognitive impairment, participated in the study. It was a 17-week feasibility study in which we used a mixed-methods approach to collect qualitative and quantitative evidence. The study included participants' recruitment, baseline, intervention, and postintervention phases. Half of the participants were randomly allocated to the treatment group (n=8), and the other half was assigned to the control group (n=8). Research assistants measured medication adherence weekly through the pill counting technique. Qualitative evidence about the system's adoption was collected through semi-structured interviews. Participants of the treatment group were interviewed regarding the system's functionalities that they perceived as most useful, less useful, and the difficulties faced while using it.

DETAILED DESCRIPTION:
1. Introduction

   One of the most common reasons for medication nonadherence among older adults is forgetfulness. Medication management technologies can help them not only with forgetfulness or cognitive impairment but also with other reasons that contribute to the lack of adherence to medications, such as polypharmacy (ie, the self-administration of multiple drugs). Research has also shown that the use of external cues supports the automatic recovery of a planned action. Therefore, this study proposes to support external cues through a tablet-based ambient display designed to increase the retrieval process of the planned action (ie, taking medications) and to provide awareness of adherence behavior. To reach this end, the Medication Ambient Display (MAD) was developed.

   An ambient display unobtrusively presents relevant information unless it requires the users' attention. In addition, users can easily monitor the display to obtain the desired information because it uses abstract modalities to represent information, such as pictures, sounds, and movement. Thus, different abstract modalities to provide external cues that enable older adults to easily obtain relevant information to take their medications on time and be aware of their medication adherence.

   MAD was implemented for Android tablets to be placed as portrait frames in the older adults' homes and to provide the following external cues:
   * Abstract and stylized representations of their medication adherence
   * Auditory and visual reminders to call older adults' attention
   * Events that may enhance older adults' awareness about whether the medication was taken.

   In this study, the effect of the use of the above-mentioned approach was assessed by using objective medication adherence measures. Moreover, qualitative findings were obtained about the adoption of the MAD.
2. Study flow

2.a. Participant recruitment

For recruiting participants, research assistants (students of the Nursing Faculty) contacted older adults affiliated in the Comunity Center of the University, in which students and academic personnel offer older adults social and health-care services. To recruit participants, research assistants administered a set of instruments to assess which older adults met the eligibility criteria. The instruments used were the Short Portable Mental State Questionnaire, the Medication Management Instrument for Deficiencies in the Elderly, and the 8-item Medication Adherence Questionnaire, also known as Morisky scale. Relatives of older adults were interviewed to identify their role in helping older adults follow their medication routine. Older adults who met the eligibility criteria and expressed their interest to participate were enrolled in the study. The recruitment procedure lasted approximately 5 weeks (weeks 1-5).

2.b. Pre-Intervention activities

Baseline data were collected during weeks 6 to 10 on medication adherence by using the pill counting technique. Research assistants noticed that participants accumulated containers with the same medications. Under those circumstances, seniors were provided with a basket to arrange the medications that should be taken each week, which facilitated data collection for measuring the Dosage_pill adherence outcome.

2.c. Intervention activities

Research assistants made a random and blind allocation of the participants to the treatment group (TG) and the control group (CG). On the first day of the intervention phase, research assistants visited older adults in the TG to introduce the MAD in the presence of caregivers by using the spaced retrieval approach, that is, teach, ask, wait, ask again, wait, and ask again. After the completion of the training session, which lasted 40 minutes approximately, the MAD was personalized according to the participant's prescriptions and through discussions with the participants on an appropriate schedule for presenting the reminders. Afterward, the MAD was placed in the area of participants' homes where they usually reported taking medications, mostly the kitchen, living room, and bedroom. The intervention phase lasted 5 weeks, during which research assistants visited participants to collect data on medication adherence (from both the TG and the CG) and system adoption (from the TG).

2.d. Postintervention activities

After the intervention was completed, MAD was removed from the participants' homes. Research assistants then carried out weekly visits (weeks 16-17) to older adults from the TG to collect data through semi-structured interviews about how MAD affected their medication routine and adherence.

3. Outcome measures and data acquisition

A set of variables were identified as relevant for analyzing the effect of the external cues provided by the MAD on the participants' medication adherence, such as dosage and timely variables, which were used to address research question 1.

During the intervention phase, qualitative evidence about the system's adoption was collected to address research question 2. The interview included questions regarding the system's functionalities that the TG's participants perceived as most useful, less useful, and the difficulties faced while using it. Similarly, at the end of the postintervention stage, TG's participants were interviewed to obtain their perceptions of how withdrawal from the MAD impacted their medication adherence. In addition, caregivers were interviewed to obtain information on their involvement in the seniors' medication activities. The questions centered on the specific activities associated with the older adults' medication regimens that caregivers were involved in and how they knew if older adults took their pills in a given week.

4. Data analysis

Student t tests and chi-square tests were used to measure the statistical difference in age, the number of prescribed medicines, and self-reported medication adherence between the TG and the CG. A one-way repeated measure analysis of variance (ANOVA), dependent t tests, and independent t tests were used to find significant differences in medication adherence between the study phases and between the TG and the CG. The McNemar test was used to verify differences within the TG between the self-reported medication adherence in the recruitment and intervention phases. To determine whether any of the differences between the means estimated are statistically significant, the P value was compared with a significance level set to .05.

For the qualitative analysis, the collected data were transcribed from their original Spanish version, that is, audio and handwritten notes. The thematic analysis approach was followed which consists of generating initial codes from the data, searching for potential themes, contrasting the identified themes with the data, and iteratively refining them.

ELIGIBILITY:
Inclusion Criteria:

* be older than 60 years
* take at least three medications prescribed by a physician (ie, polypharmacy),
* have mild cognitive impairment
* report medication-forgetting events,
* live with a relative who could report the assistance required by the study participants to take their medications.

Exclusion Criteria:

* being unable to self-administer medications due to a functionality problem or severe cognitive impairment,
* not taking pill-based medications (it may be difficult to assess adherence otherwise).

To participate in the study, it was not a requirement that older adults have experience in the use of the internet or mobile devices.

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-08-25 (Actual); Primary Completion 2017-12-08 (Actual); Study Completion 2017-12-22 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Dosage_pill | 5-week period for baseline
  It measures whether the medication is not being taken as prescribed before using MAD. It is the result of dividing the number of pills taken by participants in a period by the number of pills expected to be taken for that period. To assess the dosage_pill, research assistants collected data weekly from each participant through the pill counting technique. It was estimated for each group (TG and CG).
Change from Intervention Dosage_pill | 5-week period for intervention
  It measures whether the medication is not being taken as prescribed during the use of MAD. It is the result of dividing the number of pills taken by participants in a period by the number of pills expected to be taken for that period. To assess the dosage_pill, research assistants collected data weekly from each participant through the pill counting technique. It was estimated for each group (TG and CG).
Change from Post-Intervention Dosage_pill | 2-week period after withdrawal of MAD
  It measures whether the medication is not being taken as prescribed after the withdrawal of MAD. It is the result of dividing the number of pills taken by participants in a period by the number of pills expected to be taken for that period. To assess the dosage_pill, research assistants collected data weekly from each participant through the pill counting technique. It was estimated for TG.

SECONDARY OUTCOMES:
Dosage_MAD | 5-week period for intervention
  It is the number of medication episodes reported as taken by participants in a period divided by the number of episodes expected to be recorded for that period.
Timely | 5-week period for intervention
  It indicates whether the medication was taken in a time window (ie, 30 min) before or after the time expected to take the medication. This is the number of medication episodes registered during a period as taken in the pre-defined time window divided by the total number of medication episodes registered for that period. It was obtained for the TG.
Baseline Self-reported medication adherence | Once, in the last day of baseline period
  It is a score estimated through the 8-item Medication Adherence Questionnaire to identify participants' perception about their medication adherence. Minimum value is 0, and maximum value is 8. Higher scores mean a worse outcome (i.e., a lower medication adherence).
Change from Intervention Self-reported medication adherence | Once, in the last day of the intervention period
  It is a score estimated through the 8-item Medication Adherence Questionnaire to identify participants' perception about their medication adherence. Minimum value is 0, and maximum value is 8. Higher scores mean a worse outcome (i.e., a lower medication adherence).

CONTACTS AND LOCATIONS:
Overall Officials: Marcela D. Rodriguez, PhD, Principal Investigator — Universidad Autonoma de Baja California
Locations (1):
- Universidad Autonoma de Baja California, Mexicali, B.C., Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lavsa SM, Holzworth A, Ansani NT. Selection of a validated scale for measuring medication adherence. J Am Pharm Assoc (2003). 2011 Jan-Feb;51(1):90-4. doi: 10.1331/JAPhA.2011.09154. PMID 21247831
- [Background] Insel KC, Einstein GO, Morrow DG, Koerner KM, Hepworth JT. Multifaceted Prospective Memory Intervention to Improve Medication Adherence. J Am Geriatr Soc. 2016 Mar;64(3):561-8. doi: 10.1111/jgs.14032. PMID 27000329
- [Background] García-Vázquez, J.P., Rodríguez, M.D., Andrade, Á.G. et al. Personal and Ubiquitous Computing Journal 15(4): 389-397, 2011. https://doi.org/10.1007/s00779-010-0362-0
- [Background] Cramer JA, Roy A, Burrell A, Fairchild CJ, Fuldeore MJ, Ollendorf DA, Wong PK. Medication compliance and persistence: terminology and definitions. Value Health. 2008 Jan-Feb;11(1):44-7. doi: 10.1111/j.1524-4733.2007.00213.x. PMID 18237359
- [Background] Martinez de la Iglesia J, Duenas Herrero R, Onis Vilches MC, Aguado Taberne C, Albert Colomer C, Luque Luque R. [Spanish language adaptation and validation of the Pfeiffer's questionnaire (SPMSQ) to detect cognitive deterioration in people over 65 years of age]. Med Clin (Barc). 2001 Jun 30;117(4):129-34. doi: 10.1016/s0025-7753(01)72040-4. Spanish. PMID 11472684
- [Background] Orwig D, Brandt N, Gruber-Baldini AL. Medication management assessment for older adults in the community. Gerontologist. 2006 Oct;46(5):661-8. doi: 10.1093/geront/46.5.661. PMID 17050757
- [Derived] Zarate-Bravo E, Garcia-Vazquez JP, Torres-Cervantes E, Ponce G, Andrade AG, Valenzuela-Beltran M, Rodriguez MD. Supporting the Medication Adherence of Older Mexican Adults Through External Cues Provided With Ambient Displays: Feasibility Randomized Controlled Trial. JMIR Mhealth Uhealth. 2020 Mar 2;8(3):e14680. doi: 10.2196/14680. PMID 32130164